CLINICAL TRIAL: NCT03464864
Title: A Phase 1, Single-center, Open-label, Dose-Rising Clinical Trial to Evaluate the Pharmacokinetics, Safety and Tolerability of Treprostinil Inhalation Powder (TrIP) in Healthy Normal Volunteers
Brief Title: Pharmacokinetics, Safety and Tolerability of Treprostinil Inhalation Powder in Healthy Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MKC-475-001
Record Dates: First submitted 2018-03-01; First posted 2018-03-14 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Treprostinil Inhalation Powder 30 mcg (Experimental)
  Interventions: Drug: Treprostinil Inhalation Powder
- Treprostinil Inhalation Powder 60 mcg (Experimental)
  Interventions: Drug: Treprostinil Inhalation Powder
- Treprostinil Inhalation Powder 90 mcg (Experimental)
  Interventions: Drug: Treprostinil Inhalation Powder
- Treprostinil Inhalation Powder 120 mcg (Experimental)
  Interventions: Drug: Treprostinil Inhalation Powder
- Treprostinil Inhalation Powder 150 mcg (Experimental)
  Interventions: Drug: Treprostinil Inhalation Powder
- Treprostinil Inhalation Powder 180 mcg (Experimental)
  Interventions: Drug: Treprostinil Inhalation Powder
- Treprostinil Inhalation Powder 240 mcg (Experimental)
  Interventions: Drug: Treprostinil Inhalation Powder
- Treprostinil Inhalation Powder 300 mcg (Experimental)
  Interventions: Drug: Treprostinil Inhalation Powder

INTERVENTIONS:
Drug: Treprostinil Inhalation Powder — Single ascending dose

SUMMARY:
A Dose-Rising Clinical Trial to Evaluate the Pharmacokinetics, Safety and Tolerability of Treprostinil Inhalation Powder in Healthy Normal Volunteers

DETAILED DESCRIPTION:
Up to 48 subjects will be enrolled in 8 cohorts of 6 subjects each. The treatments are intended to establish the maximum tolerated dose in healthy normal volunteers, starting at 30 mcg. Each subject will receive one dose of Treprostinil Inhalation Powder by oral inhalation during the treatment period.

A total of 12 pharmacokinetic blood samples will be collected from each subject. Plasma pharmacokinetic samples will be analyzed for treprostinil.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily consents to participate in this study and provides written informed consent prior to the start of any study-specific procedures.
2. Male or female. Females must not be pregnant or breastfeeding.
3. Is between 18 and 55 years of age (inclusive).
4. Female subjects must weigh between 55 and 100 kg, inclusive, with a body mass index (BMI) between 19.0-32.0 kg/m2, inclusive. Male subjects must weigh between 55 and 120 kg, inclusive, with a BMI between 19.0-32.0 kg/m2, inclusive.
5. Females must be of non-childbearing potential (defined as surgically sterile [i.e. had a bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months prior to the first dose of study medication] or postmenopausal for at least 1 year prior to the first dose of study medication) or agree to use an acceptable form of birth control (see Section 4.4) from screening until 14 days after study completion.
6. Medical history, physical examination, oropharyngeal examination, vital signs, ECG, spirometry, and clinical laboratory results within normal limits or considered not clinically significant by the Investigator at screening.

Exclusion Criteria:

1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
2. A clinically significant abnormal finding on the physical exam, medical history, electrocardiogram (ECG), or clinical laboratory results at screening.
3. History of chronic lung disease such as asthma, chronic obstructive pulmonary disease (COPD), cystic fibrosis, interstitial lung disease, pulmonary fibrosis, etc.
4. History of migraine headaches.
5. History of a bleeding abnormalities (i.e., gingival bleeding, epistaxis, or blood on toilet paper, etc.) that is judged to be significant by the Investigator.
6. Has forced expiratory volume in 1 second (FEV1)/ forced vital capacity (FVC) ratio < 80% predicted or FEV25-75 <50% predicted.
7. History of anaphylaxis, a documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug.
8. Has been on a significantly abnormal diet (as determined by the Investigator) during the 4 weeks preceding the first dose of study medication.
9. Has participated in another clinical trial (and received an investigational product) within 30 days prior to the first dose of study medication.
10. Use of any over-the-counter (OTC) medication (including nutritional or dietary supplements, herbal preparations, or vitamins) within 7 days prior to the first dose of study medication until the end of study visit without evaluation and approval by the Medical Monitor.
11. Use of any prescription medication, except hormonal contraceptive or hormonal replacement therapy, from 14 days prior to the first dose of study medication until the end-of-study visit without evaluation and approval by the Investigator.
12. Has been treated with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine) within 30 days prior to the first dose of study medication, and that, in the Investigator's judgment, may impact subject safety or the validity of the study results.
13. Blood or plasma donation within 30 days prior to the first dose of study medication.
14. Smoking or use of tobacco- or nicotine-containing products within 6 months prior to the first dose of study medication until the end-of-study visit.
15. Engagement in strenuous exercise within 48 hours prior to the first dose of study medication.
16. Consumption of beverages or foods that contain alcohol, grapefruit, poppy seeds, broccoli, Brussels sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours prior to the first dose of study medication until the end-of-study visit. Subjects will be instructed not to consume any of the above products; however, allowance for an isolated single incidental consumption may be evaluated and approved by the study Investigator based on the potential for interaction with the study drug.
17. Has any prior history of substance abuse or treatment (including alcohol).
18. Is a female with a positive pregnancy test result or who is breastfeeding.
19. Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates) or cotinine.
20. Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection.
21. Unwilling to remove any artificial nails (e.g. acrylic, gel) or fingernail polish and to not use such products for the duration of the study.
22. Inability to perform study procedures including pulmonary function testing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-related adverse events (safety and tolerability) of single ascending doses of Treprostinil Inhalation Powder | At protocol-specified time points from the time of screening (day 0) to end of study (day 6)
  Incidence and severity of treatment-related adverse events determined by changes from screening (baseline) of findings from physical examinations, laboratory evaluations, vital signs measurements, pulmonary testing, and ECG measurements.

SECONDARY OUTCOMES:
Systemic exposure and pharmacokinetics of treprostinil administered as Treprostinil Inhalation Powder in healthy normal volunteers | At protocol-specified time points throughout day 1
  Concentration of treprostinil in blood as measured by protocol-specified pharmacokinetic parameters (eg maximum concentration, time to maximum concentration).
Dose proportionality | 10 months
  Dose proportionality of increasing doses of Treprostinil Inhalation Powder in healthy normal volunteers as measured by maximum blood concentration of treprostinil.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Clinical Pharmacology, Study Director — Mannkind Corporation
Locations (1):
- Investigational Site 441, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided